CLINICAL TRIAL: NCT04206371
Title: Longitudinal Follow-up of Patients With Defibrillator Threshold Testing During Implantable Cardioverter Defibrillator (ICD) Replacement
Brief Title: Defibrillation Testing During Implantable Cardioverter Defibrillator (ICD) Replacement
Acronym: T-DEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019/08
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Implantable Cardioverter-Defibrillators
Keywords: Defibrillation threshold testing; Defibrillation lead; Defibrillator replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Defibrillation testing during ICD replacment (Other)
  Interventions: Diagnostic Test: Defibrillator threshold testing

INTERVENTIONS:
Diagnostic Test: Defibrillator threshold testing — Under general or local anesthesia. Induction of Ventricular Fibrillation or R-wave synchronized shock

SUMMARY:
This study will evaluate safety and clinical outcomes of a systematic defibrillation threshold testing in patient with indication for defibrillator replacement.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillators (ICD) are strongly recommended in patients with left ventricular systolic function ≤35% or selected patients with channelopathies and cardiomyopathies.

Defibrillation threshold testing (DFT) defines the minimal energy required to successfully terminate a ventricular arrhythmia by an ICD. It remains the gold standard to evaluate the electrical integrity of the device. However inherent complications of this procedure have been registered, such as refractory ventricular fibrillation, and the need for this practice during implant and/or replacement of ICD has recently been questioned.

If several studies have led to abandonment of the DFT during initial ICD implant, its interest during replacement is still controversial. Indeed, the leads essential for the device electrical integrity are older, more fragile, and the ICD replacement may damage it.

Device replacement is indicated when battery reaches the point of Elective Replacement Interval (ERI).

Patients over 18 years old with indication for replacement of defibrillator will be included. Patient's informations (comorbidities, medical history and events during hospitalization or follow-up) and device characteristics will be collected. Procedure will be realized under local or general anesthesia and prophylactic antibiotic will be administrated. Leads will be tested before and after the implantation of the new device. After connexion of the new implanted device to the leads a DFT will be performed. Protocol of DFT will be decided by the physician who will chose between induction of ventricular fibrillation or R-wave synchronized shock. Patients will be followed for 6 and 12 months from the date of defibrillator replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ICD (VR or DR) or CRT-D undergoing generator replacement.
* Consent for participation
* Affiliation to the French social security system

Exclusion Criteria:

* Atrial Fibrillation without effective anti-coagulation treatments.
* Severe Aortic valve stenosis
* Stroke occurred in the previous month
* Hemodynamic instability contraindicating the high energy shock
* Contraindication for anesthesia
* Pregnant or breastfeeding women
* Communication difficulties or neuropsychiatric disorder
* Patients under protection of the adults (guardianship, curators or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Rate of defibrillator electrical integrity dysfunction during generator replacement. | 4 hours
  Abnormal shock impedance value.

SECONDARY OUTCOMES:
Rate of lead malfunction | 12 months
  abnormal impedance value

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Hôpital Trousseau, Chambray-lès-Tours, Centre-Val de Loire
  - Institut Lorrain du Coeur et des Vaisseaux Louis Mathieu-CHU de Nancy-Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Grand Est
  - CHU de Caen, Caen, Normandy
  - CHU de Toulouse-Hôpital Rangueil, Toulouse, Occitanie
  - Hôpital Privé du Confluent, Nantes, Pays de la Loire Region
  - Centre Hospitalier Henri Duffaut, Avignon, Provence-Alpes-Côte d'Azur Region
  - CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No